CLINICAL TRIAL: NCT03799978
Title: A Single-center, Open-label, Randomized, Two Way Crossover Study to Investigate the Food Effect on the Pharmacokinetics of ACT-541468 in Healthy Male Subjects
Brief Title: A Clinical Study to Investigate the Food Effect on the Pharmacokinetics of ACT-541468 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ID-078-113
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: Two way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: ACT-541468 50 mg under fasted conditions (Experimental): Single oral dose administered on Day 1 under fasted conditions.
  Interventions: Drug: ACT-541468
- Treatment B: ACT-541468 50 mg under fed conditions (Experimental): Single oral dose administered on Day 1 administered after food intake.
  Interventions: Drug: ACT-541468

INTERVENTIONS:
Drug: ACT-541468 — ACT-541468 50 mg film-coated tablets

SUMMARY:
This is a single-center, open-label, randomized, two way crossover study to investigate the food effect on the pharmacokinetics of ACT-541468 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* Healthy male subjects aged between 18 and 45 years (inclusive) at Screening
* Body mass index (BMI) of 18.0 to 28.0 kg/m2 (inclusive) at Screening
* No clinically relevant findings on the physical examination at Screening

Exclusion Criteria:

* History of major medical or surgical disorders, which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatments (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol
* Modified Swiss Narcolepsy Scale total score < 0 at screening or history of narcolepsy or cataplexy

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic endpoint: AUC0-24 | Multiple timepoints; duration: up to 48 hours in each treatment period
  Area under the plasma concentration-time curve (AUC) from time zero to 24 h

OTHER OUTCOMES:
Pharmacokinetic endpoint: AUC0-inf | Multiple timepoints; duration: up to 48 hours in each treatment period
  AUC from time zero to infinity
Pharmacokinetic endpoint: Cmax | Multiple timepoints; duration: up to 48 hours in each treatment period
  Maximum plasma concentration
Pharmacokinetic endpoint: tmax | Multiple timepoints; duration: up to 48 hours in each treatment period
  Time to reach maximum plasma concentration
Pharmacokinetic endpoint: t½ | Multiple timepoints; duration: up to 48 hours in each treatment period
  Terminal elimination half-life
Treatment-emergent adverse events | From study treatment administration up to EOT; duration: up to 48 hours in each treatment period
Serious treatment-emergent adverse events | From study treatment administration up to EOT; duration: up to 48 hours in each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CEPHA s.r.o., Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No